CLINICAL TRIAL: NCT00571376
Title: Evaluating the Impact on Quality and Costs of Regional Clinical Data Exchange Programs in New York State
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The Commonwealth Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 20060550
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Quality of Health Care; Health Care Costs
Keywords: Quality of health care; Health care costs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Those exposed to health information technology or health information exchange
  Interventions: Other: Health information technology and exchange
- 2: Those not exposed to health information technology or health information exchange

INTERVENTIONS:
Other: Health information technology and exchange — Health information technology includes electronic health records, electronic prescribing, and electronic results notification and/or viewers. Health information exchange includes use of central repositories of data and peer-to-peer models.
  Groups: 1

SUMMARY:
The purpose of this study is to measure the financial effects of health information technology and health information exchange in regional health information organizations in New York State.

DETAILED DESCRIPTION:
In 2004, the federal government set an ambitious goal of ensuring that most Americans have electronic health records within 10 years and the presence of a widespread clinical information exchange capability will greatly facilitate this goal. Through HEAL NY, New York State is currently awarding millions of dollars in grants to support health information technology initiatives across the state through regional clinical information exchanges. The financial success of these initiatives is expected to result from improvements in health care quality and efficiency. However, whether these initiatives will be cost saving, as experts assert, and what the return-on-investments of these initiatives will be are unknown. Answering these questions will provide critical information to the nation as we progress towards a national health information network. We will conduct a multi-center financial evaluation of regional clinical information exchanges. The results of the financial evaluations proposed in this study will provide a framework and standardized methodology including metrics for financial evaluations of regional health information organizations and return-on-investment analyses from the perspectives of providers and payers. We will consider the financial effects as driven by changes in quality, safety, and efficiency.

The most advanced community we studied was Rochester, NY, and studying this community allowed us to measure the effects of health information technology and health information exchange on 3 major utilization outcomes (hospital admissions, hospital re-admissions, and repeat medical imaging).

ELIGIBILITY:
Inclusion Criteria:

* Patients and health care providers participating in regional health information organizations or their affiliate institutions.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and health care providers in the Rochester, NY community
Sampling Method: Non-Probability Sample
Enrollment: 218766 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hospital admissions | 2 years
Hospital re-admissions | 2 years
Repeat medical imaging | 2 years

SECONDARY OUTCOMES:
Usage of health information technology and health information exchange | 2 years
Changes in health care quality | 2 years
Changes in patient safety | 2 years
Changes in health care efficiency | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rainu Kaushal, MD, MPH, Principal Investigator — Weill Medical College of Cornell University; Lisa M Kern, MD, MPH, Study Director — Weill Medical College of Cornell University
Locations (1):
- Rochester RHIO, Rochester, New York, United States